CLINICAL TRIAL: NCT06296602
Title: Screening Anal HPV Colonization in Men Sex Men Using Pre-exposure Prophylaxis for HIV
Brief Title: Screening Anal HPV Colonization in Men Sex Men Using Pre-exposure Prophylaxis for HIV (ANAPreP'HPV)
Acronym: ANAPreP'HPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023/777
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: PreP

STUDY DESIGN:
Intervention Model Description: A prelevement for HPV genotyping and anal cytology will be carried out in addition to the anal swabs taken quarterly to screen for other sexually transmitted infections.
  A questionnaire will be completed by the doctor to record the data of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANAPreP-HPV (Experimental): A prelevement for HPV genotyping and anal cytology will be carried out in addition to the anal swabs taken quarterly to screen for other sexually transmitted infections.
  A questionnaire will be completed by the doctor to record the data of interest.
  Interventions: Other: A prelevement for HPV genotyping and anal cytology will be carried out in addition to the anal swabs taken quarterly to screen for other sexually transmitted infections.

INTERVENTIONS:
Other: A prelevement for HPV genotyping and anal cytology will be carried out in addition to the anal swabs taken quarterly to screen for other sexually transmitted infections. — A prelevement for HPV genotyping and anal cytology will be carried out in addition to the anal swabs taken quarterly to screen for other sexually transmitted infections. A questionnaire will be completed by the doctor to record the data of interest.
  Other Names: A questionnaire will be completed by the doctor to record the data of interest

SUMMARY:
This is an interventional study investigating HPV carriage and liquid-based cytology at anal level. It will be offered to all patients undergoing PreP consultations at Besançon University Hospital. The anal swab will be taken by the doctor using a cyto-brush during the consultation.

DETAILED DESCRIPTION:
The duration of participation in the study is 3 months for the submission of the results of the samples. A medical proctology consultation may also be offered, depending on the results of the screening.

This will be carried out in addition to the anal swabs taken quarterly to screen for other sexually transmitted infections.

A questionnaire will be completed by the doctor to record the data of interest. From additional data already entered in the e-NADIS software will be included for study.

ELIGIBILITY:
Inclusion Criteria:

Men sex Men Using Pre-exposure Prophylaxis for HIV Follow up au CHU de Besançon.

Exclusion Criteria:

* Women
* No MSM
* Under 18
* History of HPV related cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-11-04 (Estimated); Study Completion 2024-11-04 (Estimated)

PRIMARY OUTCOMES:
prevalence HPV | day 1
  prevalence HPV
typing HPV | day 1
  typing HPV

SECONDARY OUTCOMES:
High risk HPV risk factors | day 1
  High risk HPV risk factors
Cytologist abnormalies | day 1
  Cytologist abnormalies

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No